CLINICAL TRIAL: NCT03679728
Title: Sensorimotor Outcomes of Children Exposed to Foetal Zika Virus Infection During the First or Second Trimester of Gestation.
Brief Title: Sensorimotor Outcomes of Children Exposed to Foetal Zika Virus Infection
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Carlos Bandeira de Mello Monteiro, Associate Professor, University of Sao Paulo
Other Study IDs: 65822017.3.0000.5390
Record Dates: First submitted 2018-09-16; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Zika Virus Infection
Keywords: Zika virus; Children; Microcephaly
MeSH Terms: conditions — Zika Virus Infection; Microcephaly | interventions — Pregnancy Trimester, First; Pregnancy Trimester, Second

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First trimester: Group of children from mother affected by Zika virus in the first trimester of pregnancy.
  Interventions: Behavioral: First trimester
- Second trimester: Group of Children from mother affected by Zika virus in the second trimester of pregnancy.
  Interventions: Behavioral: Second trimester

INTERVENTIONS:
Behavioral: First trimester — Analysis of sensorimotor outcomes
  Groups: First trimester
Behavioral: Second trimester — Analysis of sensorimotor outcomes
  Groups: Second trimester

SUMMARY:
Introduction: It is estimated that more than one million Brazilians were infected by zika virus in the last two years. Brazilian researchers first noted the virus's potential association with microcephaly. Objective: This study aimed to describe the motor performance of children aged between 6-18 months with the diagnoses of congenital Zika syndrome. Method: This is a cross-sectional, prospective and descriptive study. The study population consisted of 31 children. Participants were evaluated using Alberta Infant Motor Scale (AIMS) and Gross Motor Function Measure (GMFM).

DETAILED DESCRIPTION:
Method This was a cross-sectional, prospective and descriptive study. This study was approved by the Ethics Committee for Analysis of Research Projects of the University of São Paulo - School of Arts, Sciences and Humanities - EACH, under the protocol number approved CAAE: 65822017.3.0000.5390. Parents or caregivers gave written informed consent prior to participating. Children were evaluated by Physiotherapists who had at least two years of neuropediatric practice in the cities of Arcoverde and Recife in Pernambuco, Brazil.

Sample Participants were evaluated in Salud Serviços de Reabilitação Clinic (Recife) and Mens Sana Clinic (Arcoverde) using Alberta Infant Motor Scale (AIMS - prone, supine, sitting, standing, total score and corresponding percentile) and Gross Motor Function Measure (GMFM, A: lying/rolling and B: sitting). Head circumference at birth and on the day of assessment (in cm), age (in months) and family income, as well as AIMS and GMFM scores, provided as means, standard deviations, and minimum and maximum scores. Qualitative data about sex, muscle tone (increased, decreased or normal), visual/ hearing impairments (yes or no) were also collected.

Assessment Scales To assess performance of the children the following motor scales and assessments were used.

1. Alberta Infant Motor Scale (AIMS) is a reliable and easy-to-use clinical assessment tool for the evaluation of infant gross motor development from birth until the acquisition of independent walking. AIMS is a norm-referenced measure of infant gross motor development. It contains 58 items, which assess the control and integrity of the antigravity muscles during observation of infant motor skills in prone, supine, sitting, and standing positions. It has been recognized as a useful tool to assess gross motor maturation during infancy, to trace motor delay, and to identify infants who may benefit from early intervention Supine, prone, sitting, standing scores and the total score were registered, as well as the age corresponding percentiles. Interpretation of an AIMS score is never made at the level of individual items, rather it is derived from percentile ranking established through plotting an infant's age to the closest week and his or her total score on the centile graph, the percentile rankings provided on the centile graph would be unaffected for all infants because all age differences are less than one week.
2. The Gross Motor Function Measure (GMFM) is a clinical tool designed to evaluate the change in gross motor function in children with disabilities. This measure consists of 88 items that evaluate lying and rolling up to walking, running and jumping skills. There is a four-point scoring system for each item on the GMFM and can be used with children above 6 months. In the present study, only dimensions A (lying and rolling) and B (sitting) were used. Item scores can be summed to calculate raw and percentile scores for each of the GMFM dimensions, selected goal areas and a total score.

ELIGIBILITY:
Inclusion Criteria:

* birth weight between 2,000 and 4,000 g,
* gestational age between 35 and 42 weeks,
* zika maternal infection (confirmed by blood or urine exam) in the first or second gestation trimesters and having head circumference below 33 cm at birth.

Exclusion Criteria:

* Other diseases or injuries at birth such as Traumatic brain injury,
* Parenchymal hemorrhage,
* Hypoxic Ischemic Encephalopathy (HIE),
* Obstetric brachial palsy.

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consisted of 31 children from mother affected with Zika Virus, in Arcoverde and Recife in Pernambuco, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2017-04-16 (Actual)

PRIMARY OUTCOMES:
Children with microcephaly at birth, whose mothers had zika virus infection in the first or second gestation trimester, showed poor sensorimotor outcomes, mainly impaired muscle tone and antigravity postural control. | 1 month
  Sensorimotor outcomes was assessed by using Alberta Infant Motor Scale (AIMS)

SECONDARY OUTCOMES:
Children whose mothers were affected in the first trimester had lower head circumference measures that children whose mothers were affected in the second trimester. | 1 month
  Assessment of birth head circumference.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos BM Monteiro, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Arts, Sciences and Humanities of the University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided